CLINICAL TRIAL: NCT02535234
Title: Comparison of the Subjective and Objective Performance of a Novel Continuous Positive Airway Pressure (CPAP) System With a Traditional Continuous Positive Airway Pressure (CPAP) System.
Brief Title: Comparison of Two Continuous Positive Airway Pressure Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MA011015
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnoea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Participants randomised to Arm 1 will receive an intervention of 7 nights with the Novel system followed by 7 nights with theTraditional system
  Interventions: Device: Novel System; Device: Traditional System
- Arm 2 (Active Comparator): Participants randomised to Arm 1 will receive an intervention of 7 nights with the Traditional system followed by 7 nights with the Novel system
  Interventions: Device: Novel System; Device: Traditional System

INTERVENTIONS:
Device: Novel System — A Novel full Continuous Positive Airway Pressure (CPAP) system - Prototype Device, Mask + Accessories
Device: Traditional System — A Traditional full Continuous Positive Airway Pressure (CPAP) system- Released Device + Accessories, Prototype Mask
  Other Names: AirSense System

SUMMARY:
Randomised crossover trial of a novel and traditional Continuous Positive Airway Pressure (CPAP) system in Obstructive Sleep Apnoea patients.

ELIGIBILITY:
Inclusion Criteria

* Participant is willing to provide written informed consent
* Participant is able to read and comprehend written and spoken English
* Participant is ≥ 18 years of age
* Participant has been diagnosed with Obstructive Sleep Apnoea (OSA)
* Participants has been established on Continuous Positive Airway Pressure (CPAP) for ≥ 6 months
* Participants is currently using the same mask type/variant as the interventional mask system to be evaluated
* Participants is able to participate for the duration of the study

Exclusion Criteria

* Participant is not willing to provide written informed consent
* Participant is unable to read and comprehend written and spoken English
* Participant is < 18 years of age
* Participant has not been diagnosed with Obstructive Sleep Apnoea (OSA)
* Participant has not been established on Continuous Positive Airway Pressure (CPAP) for ≥ 6 months
* Participant is not currently using the same mask type/variant as the interventional mask system to be evaluated
* Participant is unable to participate for the duration of the study
* Participant is pregnant
* Participant is established on bi-level support therapy
* Participant, or participants bed partner, has metallic implants in head neck or chest
* Participant has a with a pre-existing lung disease or a condition that would predispose them to pneumothorax (e.g. Chronic Obstructive Pulmonary Disease (COPD), lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection, lung injury)
* Participant is unsuitable to participate in the study in the opinion of the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Subjective usability ratings of the prototype system using a visual analogue scale, compared to a reference level and the second full system. | 1 year
  Participants will be asked to complete a short questionnaire at the end of each week to evaluate the general usability of the system. The questionnaire will include questions related to system use and comfort. The participants will answer the questions using an 11-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, Principal Investigator — ResMed Limited; Holger Woehrle, MD, Principal Investigator — ResMed
Locations (1):
- ResMed, Sydney, New South Wales, Australia

REFERENCES:
- [Result] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Result] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Result] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871